CLINICAL TRIAL: NCT03058276
Title: New Therapeutic Strategies for Inhibitory Control Improvement of Alcohol-dependent Patients
Brief Title: New Therapeutic Strategies for Inhibitory Control in Alcoholism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Principal Investigator, Gabriel Rubio Valladolid, MD, Psychiatrist, MD, PhD, Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/099
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Alcoholism
Keywords: rTMS; AAT; Alcohol-Dependence; Relapses
MeSH Terms: conditions — Alcoholism; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded experiment regarding rTMS treatment is applied to both subjects and investigators. The only non-masked role is for the technician applying either Magstim Rapid or SAM coils to each group of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exposure (Experimental): Exposure to a 5 minutes video related to alcohol consumption (updating/retrieval), followed by 10 minutes of the alcohol- AAT(Approach Avoidance Task) (extinction), during 4 days of training (2 weeks).
  Interventions: Behavioral: Retrieval-Extinction Learning
- No exposure (Active Comparator): Exposure to a 5 minutes video with neutral content (no retrieval) followed by 10 minutes of the alcohol- AAT (Approach Avoidance Task) , during 4 days of training.
  Interventions: Behavioral: Retrieval-Extinction Learning
- Active rTMS (Experimental): Each session (5 sessions along 2 weeks), patients receive active stimulation with repetitive transcraneal magnetic stimulation (rTMS) of the right dorsolateral prefrontal cortex.
  Interventions: Other: rTMS
- SAM (Sham Comparator): Pacients receiving a sham stimulation (SAM), with a similar procedure to the experimental condition
  Interventions: Other: SAM

INTERVENTIONS:
Behavioral: Retrieval-Extinction Learning — The intervention consists of the accomplishment of the task of approach-avoidance of alcohol during 4 days of training. Subjects are instructed to respond with an approach movement (pulling a lever) to neutral images and to respond with avoidance movement (pushing the lever) to images of alcohol.
  Arms: Exposure; No exposure
Other: rTMS — Previous to rTMS completion, MRI scans were performed in order to determinate the motor threshold trough 1Hz stimuli and locate the desired area with the neuronavigator. Motor threshold is defined as the stimulus with less intensity, able to generate a motor potential of at least 50 µV in 10 trials. Next, patients were called for 5 times per week, along 2 weeks, for receiving brain stimulation with Magstim Rapid coil. rTMS is performed at 10 Hz, during 4.9 seconds,for each set of stimuli (20), with a interval between sets of 30 seconds.
  Arms: Active rTMS
Other: SAM — Previous to rTMS completion, MRI scans were performed in order to determinate the motor threshold trough 1Hz stimuli and locate the desired area with the neuronavigator. Motor threshold is defined as the stimulus with less intensity, able to generate a motor potential of at least 50 µV in 10 trials. Next, patients were called for 5 times per week, along 2 weeks, for receiving brain stimulation with SAM coil.
  Arms: SAM

SUMMARY:
This experimental research studies the efficacy of two different treatments for inhibitory control improvement in alcohol-dependent individuals, one consisting of Retrieval-Extinction Learning ( alcohol AAT Task) and the other consisting in rTMS of the right dorsolateral prefrontal cortex.

DETAILED DESCRIPTION:
The main purpose of this study is to demonstrate the efficacy of two different treatments for inhibitory control improvement (measured by the modified Stop signal task): a behavioral treatment based on Retrieval-Extinction Learning, through the AAT (Alcohol Approach Avoiding Task) and a treatment based on the neuromodulation of prefrontal cortex through the rTMS (repetitive transcraneal magnetic stimulation) technique. To carry out this study, 105 alcoholic patients will be compared for clinical variables (abstinence/relapses), self-informed (UPPS) and behvavioral impulsivity (Stop signal task), along with biological measures for polymorphism determinations. Alcohol-dependent individuals will be divided into 4 groups of study (1:1 proportion for Retrieval-Extinction Learning with AAT and 2:1 (double for the effective technique comparing to placebo/control) for rTMS): Group 1 (N=30): exposure to an alcohol-related video followed by AAT; Group 2 (N=30): neutral-content video followed by AAT; Group 4 (30): active stimulation rTMS (10 Hz) ; Group 4 (N=15): placebo stimulation SAM.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 50 years old.
* A minimum of 28 days of abstinence
* Consent to participate in the study.

Exclusion Criteria:

* Subjects with other substance dependence ( with the exception of tobacco)
* Subjects with a history of brain injury or neurological diseases
* Denial for study participation
* Non-spanish speakers
* rTMS selected participants with be assed in order to discard epilepsy, presence for metallic elements and CNS valves

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Relapses | 3 months
  Number of relapses
Heavy drinking | 3 months
  Number of days of heavy drinking
Abstinence | 3 months
  Days of accumulated abstinence

SECONDARY OUTCOMES:
Behavioral Impulsivity | 2 days
  Stop signal task reaction times
Self-reported Impulsivity | 2 days
  scores for UPPS
Polymorphism distribution of CRH and ANK3 genes | 2 days
  Biological determinations-lymphocyte samples

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Rubio Valladolid, Psychiatrist, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiers RW, Eberl C, Rinck M, Becker ES, Lindenmeyer J. Retraining automatic action tendencies changes alcoholic patients' approach bias for alcohol and improves treatment outcome. Psychol Sci. 2011 Apr;22(4):490-7. doi: 10.1177/0956797611400615. Epub 2011 Mar 9. PMID 21389338
- [Background] Mishra BR, Nizamie SH, Das B, Praharaj SK. Efficacy of repetitive transcranial magnetic stimulation in alcohol dependence: a sham-controlled study. Addiction. 2010 Jan;105(1):49-55. doi: 10.1111/j.1360-0443.2009.02777.x. PMID 20078462